CLINICAL TRIAL: NCT05477186
Title: A Phase 1, Open-label, Safety and Immunogenicity Study of a Booster Dose of the Investigational CV0501 mRNA COVID-19 Vaccine in Adults at Least 18 Years Old
Brief Title: Safety and Immunogenicity Study of a Booster Dose of the Investigational CV0501 mRNA COVID-19 Vaccine in Adults at Least 18 Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 218595
Record Dates: First submitted 2022-07-27; First posted 2022-07-28 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19; Pandemic; Booster vaccination
MeSH Terms: conditions — COVID-19 | interventions — CV0501 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: CV0501 Dose Cohort 1 (12 μg) (Experimental): Healthy participants received a single dose of 12 microgram (μg) CV0501 vaccine intramuscularly at Day 1.
  Interventions: Biological: CV0501 (12 μg)
- Part A: CV0501 Dose Cohort 2 (25 μg) (Experimental): Healthy participants received a single dose of 25 μg CV0501 vaccine intramuscularly at Day 1.
  Interventions: Biological: CV0501 (25 μg)
- Part A: CV0501 Dose Cohort 3 (50 μg) (Experimental): Healthy participants received a single dose of 50 μg CV0501 vaccine intramuscularly at Day 1.
  Interventions: Biological: CV0501 (50 μg)
- Part A: CV0501 Dose Cohort 4 (100 μg) (Experimental): Healthy participants received a single dose of 100 μg CV0501 vaccine intramuscularly at Day 1.
  Interventions: Biological: CV0501 (100 μg)
- Part A: CV0501 Dose Cohort 5 (200 μg) (Experimental): Healthy participants received a single dose of 200 μg CV0501 vaccine intramuscularly at Day 1.
  Interventions: Biological: CV0501 (200 μg)
- Part B: CV0501 Dose Cohort 6 (3 μg) (Experimental): Healthy participants received a single dose of 3 μg CV0501 vaccine intramuscularly at Day 1.
  Interventions: Biological: CV0501 (6 μg)
- Part B: CV0501 Dose Cohort 7 (6 μg) (Experimental): Healthy participants received a single dose of 6 μg CV0501 vaccine intramuscularly at Day 1.
  Interventions: Biological: CV0501 (3 μg)

INTERVENTIONS:
Biological: CV0501 (3 μg) — Study vaccine was administered as a single intramuscular injection.
  Arms: Part B: CV0501 Dose Cohort 7 (6 μg)
Biological: CV0501 (6 μg) — Study vaccine was administered as a single intramuscular injection.
  Arms: Part B: CV0501 Dose Cohort 6 (3 μg)
Biological: CV0501 (12 μg) — Study vaccine was administered as a single intramuscular injection.
  Arms: Part A: CV0501 Dose Cohort 1 (12 μg)
Biological: CV0501 (25 μg) — Study vaccine was administered as a single intramuscular injection.
  Arms: Part A: CV0501 Dose Cohort 2 (25 μg)
Biological: CV0501 (50 μg) — Study vaccine was administered as a single intramuscular injection.
  Arms: Part A: CV0501 Dose Cohort 3 (50 μg)
Biological: CV0501 (100 μg) — Study vaccine was administered as a single intramuscular injection.
  Arms: Part A: CV0501 Dose Cohort 4 (100 μg)
Biological: CV0501 (200 μg) — Study vaccine was administered as a single intramuscular injection.
  Arms: Part A: CV0501 Dose Cohort 5 (200 μg)

SUMMARY:
Prevention of COVID-19 caused by SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide documented informed consent prior to any study procedures being performed
2. Is capable of understanding and agrees to comply with planned study procedures and to be available for all study visits
3. Has received at least 2 doses of Comirnaty or Moderna COVID-19 Vaccine (Spikevax®\), with the last dose of vaccine received at least 6 months prior to screening
4. Negative for SARS-CoV-2 infection by RT-PCR test at screening
5. Is a male or nonpregnant female >= 18 years old
6. If the participant is a woman of childbearing potential, the participant agrees to use at least 1 highly effective form of contraception for at least 30 days prior to the study vaccination up to 3 months after study vaccination.
7. Agrees to refrain from blood or plasma donation from the first study vaccination through end of study.
8. Has a body mass index of 18 to 40 kg/m^2, inclusive, at screening.
9. Is healthy or medically stable as determined by investigator judgment based on medical history, clinical laboratory tests, vital sign measurements, and physical examination findings

Exclusion Criteria:

1. Participant is female and has a positive pregnancy test result at screening.
2. Participant is female and is breastfeeding or will (re)start breastfeeding from the study vaccination to 3 months after vaccination.
3. Has an acute febrile illness with temperature >=38.0°C or >=100.4°F within 72 hours before study vaccination. Individuals with suspected COVID-19 symptoms should be excluded and referred for medical care.
4. Has a history of documented SARS-CoV-2 infection or COVID-19 within 6 months before screening.
5. Has a documented medical history of HIV, hepatitis B or hepatitis C infection prior to screening, or a positive test for these conditions at screening.
6. Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (eg, malignancy) or immunosuppressive/cytotoxic therapy (eg, medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders). Chronic use (more than 14 continuous days) of any medication that may be associated with changes in immune function including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy immunotherapy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar or toxic drugs within 6 months of the first study vaccination. Inclusion of persons who use low dose topical, ophthalmic, inhaled, or intranasal steroid preparations is permitted.
7. History of myocarditis, pericarditis, or idiopathic cardiomyopathy, or presence of any medical condition that increases risk of myocarditis or pericarditis, including cocaine abuse, cardiomyopathy, endomyocardial fibrosis, hypereosinophilic syndrome, hypersensitivity myocarditis, eosinophilic granulomatosis with polyangiitis, persistent myocardial viral infection (eg, due to enterovirus or adenovirus), and celiac disease.
8. Has a new onset, clinically significant, abnormal biochemistry or hematology finding (defined as >= Grade 1) at screening (adults with Grade 1 laboratory abnormalities that have been stable for at least 6 months before enrollment may be included in the study).
9. Individuals with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to: systemic or cutaneous lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, Guillain- Barré syndrome, multiple sclerosis, Sjögren's syndrome, idiopathic thrombocytopenia purpura, glomerulonephritis, autoimmune thyroiditis, giant cell arteritis (temporal arteritis), Takayasu arteritis, granulomatosis with polyangiitis, psoriasis, and insulin-dependent diabetes mellitus (Type 1).
10. Has an unstable chronic medical condition. This refers to a condition requiring a new medication or increase in dose of current medication(s) or a condition requiring hospitalization within 6 months prior to screening.
11. Has a history of hypersensitivity or severe allergic reaction, including anaphylaxis, generalized urticaria, angioedema, and other significant reactions, to vaccines or to any component of the investigational product.
12. Has received or plans to receive any licensed vaccine, within 4 weeks before or 4 weeks after study vaccination. Inactivated vaccines for influenza are permitted during the study if they are administered at least 14 days before or after study vaccination.
13. Has had known close contact with anyone who had a confirmed SARS-CoV-2 infection within 2 weeks before study vaccination. Rescreening of these participants permitted after quarantine period is complete.
14. Has participated or plans to participate in another investigational study involving any investigational product or device within 6 months or 5 half-lives, whichever is longer, before the study vaccination through end of study.
15. Has received or plans to receive immunoglobulins or any blood or blood products within 3 months before the first study vaccination through end of study.
16. Has a bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
17. Has a history of alcohol abuse or other recreational drug use (excluding cannabis) within 6 months before study vaccination.
18. Has any abnormal skin condition or permanent body art (eg, tattoo) that would interfere with the ability to observe local reactions at the injection site.
19. Has a medical disease or psychiatric condition that, in the opinion of the investigator, precludes study participation because it would place the individual at an unacceptable risk of injury, render the individual unable to meet the requirements of the protocol or interfere with the individual's successful completion of the trial.
20. Participant is an employee or family member of the investigator or study site personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (11):
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Norfolk, Virginia
- Australia (4):
  - GSK Investigational Site, Brookvale, New South Wales
  - GSK Investigational Site, Merewether, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
- Philippines (2):
  - GSK Investigational Site, Cavite
  - GSK Investigational Site, Iloilo City

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Essink BJ, Shapiro C, Isidro MGD, Bradley P, Pragalos A, Bloch M, Santiaguel J, Frias MV, Miyakis S, Alves de Mesquita M, Berre S, Servais C, Waugh N, Hoffmann C, Baba E, Schonborn-Kellenberger O, Wolz OO, Koch SD, Ganyani T, Boutet P, Mann P, Mueller SO, Ramanathan R, Gaudinski MR, Vanhoutte N. Safety and immunogenicity of a modified mRNA-lipid nanoparticle vaccine candidate against COVID-19: Results from a phase 1, dose-escalation study. Hum Vaccin Immunother. 2024 Dec 31;20(1):2408863. doi: 10.1080/21645515.2024.2408863. Epub 2024 Oct 18. PMID 39422261
- [Derived] Roth N, Gergen J, Kovacikova K, Mueller SO, Ulrich L, Schon J, Halwe NJ, Fricke C, Corleis B, Dorhoi A, Hoffmann D, Beer M, Maione D, Petsch B, Rauch S. Assessment of Immunogenicity and Efficacy of CV0501 mRNA-Based Omicron COVID-19 Vaccination in Small Animal Models. Vaccines (Basel). 2023 Jan 31;11(2):318. doi: 10.3390/vaccines11020318. PMID 36851196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 centers in Australia, Philippines and United States.
Pre-assignment Details: Escalation to the next higher dose cohorts was based on the Safety Review Team (SRT) review of safety data from the same age group.
Groups:
- Part B: CV0501 Dose Cohort 6 (3 μg): Healthy participants received a single dose of 3 microgram (μg) CV0501 vaccine intramuscularly at Day 1.
- Part A: CV0501 Dose Cohort 1 (12 μg): Healthy participants received a single dose of 12 μg CV0501 vaccine intramuscularly at Day 1.
Period: Overall Study
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg)
Started | 15 | 17 | 31 | 30 | 31 | 31 | 30
Safety Set | 15 | 15 | 30 | 30 | 30 | 30 | 30
Per Protocol Immunogenicity (PPI) | 15 | 14 | 28 | 27 | 28 | 29 | 26
Completed | 13 | 15 | 28 | 29 | 29 | 30 | 28
Not Completed | 2 | 2 | 3 | 1 | 2 | 1 | 2
Not completed — Vaccine not administered | 0 | 2 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on enrolled set which includes all participants who have a signed Informed Consent Form and were assigned to a group, vaccinated, or had an immunogenicity blood draw.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg) | Total
Number analyzed (Participants) | 15 | 17 | 31 | 30 | 31 | 31 | 30 | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (12.18) | 35.8 (12.66) | 50.9 (16.43) | 48.9 (17.99) | 54.5 (15.69) | 55.2 (16.15) | 49.8 (19.23) | 49.2 (17.37)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 11 | 7 | 7 | 11 | 13 | 11 | 18 | 78
  Female | 4 | 10 | 24 | 19 | 18 | 20 | 12 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 10 | 7 | 7 | 6 | 3 | 38
  Not Hispanic or Latino | 12 | 15 | 21 | 23 | 24 | 25 | 27 | 147
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Adverse Events (AE) During 7 Days After Vaccination
Description: Assessed solicited local adverse events were injection site pain, redness, swelling, and Lymphadenopathy.
Time Frame: From Day 1 to Day 7 (including Day 7)
Population: Analysis was performed on the Safety set who received 1 dose of investigational product. Only participants in the Safety Set with at least one day of eDiary entry within each dose group and at each level of summarization were included in this analysis; one participant in the 25 μg group did not complete the eDiary and was excluded from the summary.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg)
Number analyzed (Participants) | 15 | 15 | 30 | 29 | 30 | 30 | 30
Participants
  Overall | 5 | 9 | 16 | 19 | 16 | 19 | 22
  Injection site pain | 5 | 9 | 14 | 19 | 15 | 19 | 22
  Redness | 0 | 0 | 1 | 2 | 2 | 1 | 9
  Swelling | 1 | 1 | 0 | 1 | 3 | 1 | 6
  Lymphadenopathy | 0 | 2 | 4 | 2 | 5 | 4 | 6

2. Primary Outcome: Number of Participants With Solicited Systemic AE During 7 Days After Vaccination
Description: Assessed solicited systemic AEs were fever, headache, fatigue, myalgia, arthralgia, and chills.
Time Frame: From Day 1 to Day 7 (including Day 7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg)
Number analyzed (Participants) | 15 | 15 | 30 | 29 | 30 | 30 | 30
Participants
  Overall | 4 | 4 | 11 | 17 | 15 | 18 | 21
  Fever | 0 | 0 | 0 | 0 | 2 | 3 | 2
  Headache | 3 | 4 | 5 | 9 | 9 | 13 | 13
  Fatigue | 1 | 0 | 5 | 14 | 10 | 15 | 14
  Myalgia | 2 | 3 | 8 | 10 | 10 | 16 | 17
  Arthralgia | 0 | 1 | 2 | 5 | 3 | 6 | 3
  Chills | 1 | 0 | 3 | 5 | 3 | 11 | 11

3. Primary Outcome: Number of Participants With Unsolicited AEs for 28 Days After Study Vaccination
Description: An unsolicited AE is defined as any AE that is volunteered from the participant and occurs within 28 days after vaccination.
Time Frame: From Day 1 to day 28 (including day 28)
Population: Analysis was performed on the Safety set who received 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg)
Number analyzed (Participants) | 15 | 15 | 30 | 30 | 30 | 30 | 30
Participants | 4 | 1 | 2 | 2 | 4 | 5 | 8

4. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAEs) From Study Vaccination Through the End of the Study
Description: An MAAE is defined as an AE that results in a visit to a medical professional. Medically attended visits are defined as a telemedicine visit, physician's office visit, urgent care visit, emergency room visit, hospitalization, or death.
Time Frame: From Day 1 up to Day 180 (including Day 180)
Population: Analysis was performed on the Safety set who received 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg)
Number analyzed (Participants) | 15 | 15 | 30 | 30 | 30 | 30 | 30
Participants | 2 | 2 | 9 | 2 | 5 | 6 | 4

5. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs) From Study Vaccination Through the End of the Study
Description: An AESI (serious or nonserious) is defined as an AE or serious adverse event (SAE) of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor could be appropriate.
Time Frame: From Day 1 up to Day 180 (including Day 180)
Population: Analysis was performed on the Safety set who received 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg)
Number analyzed (Participants) | 15 | 15 | 30 | 30 | 30 | 30 | 30
Participants | 2 | 0 | 1 | 3 | 2 | 4 | 3

6. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) From Study Vaccination Through the End of the Study
Description: An SAE is defined as any event that: Results in death Is immediately life-threatening Requires inpatient hospitalization or prolongation of existing hospitalization Results in persistent or significant disability/incapacity Is a congenital anomaly/birth defect Is a spontaneous miscarriage Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered SAEs when, based upon appropriate medical judgment, they may jeopardize the participant or may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.
Time Frame: From Day 1 up to Day 180 (including Day 180)
Population: Analysis was performed on the Safety set who received 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg)
Number analyzed (Participants) | 15 | 15 | 30 | 30 | 30 | 30 | 30
Participants | 0 | 0 | 0 | 0 | 1 | 2 | 0

7. Secondary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibody (Ab) Against Pseudovirus Bearing S Protein From SARS-CoV-2 WT, Omicron, and Delta Variants at Each Collection Timepoint
Time Frame: At Day 1, Day 15, Day 29, Day 91, and Day 181
Population: The Per Protocol Immunogenicity (PPI) Set includes all eligible participants who received a dose of investigational product per protocol and who have values at specific timepoint for neutralizing Ab titers against pseudovirus bearing S protein from the Omicron variant of SARS-CoV-2.
Measure: Geometric Mean (Standard Deviation); unit: Titers
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg)
Number analyzed (Participants) | 15 | 14 | 28 | 27 | 28 | 29 | 26
Titers
  Wild Type (WT), Day 1 | 1311.5 (5.36) | 1154.5 (3.01) | 1678.3 (3.81) | 884.4 (3.67) | 1752.1 (3.25) | 1248.6 (4.14) | 1556.0 (4.83)
  WT, Day 15: number analyzed (Participants) | 13 | 14 | 27 | 27 | 25 | 24 | 24
  WT, Day 15 | 3478.1 (2.67) | 3663.7 (2.04) | 7344.4 (2.22) | 4651.9 (2.44) | 9679.4 (2.19) | 11321.4 (2.01) | 20966.2 (2.49)
  WT, Day 29: number analyzed (Participants) | 13 | 14 | 27 | 26 | 26 | 26 | 21
  WT, Day 29 | 3065.6 (2.66) | 2865.2 (2.59) | 6188.1 (2.25) | 5869.7 (2.64) | 12148.6 (2.42) | 8356.7 (2.36) | 15717.3 (2.62)
  WT, Day 91: number analyzed (Participants) | 10 | 14 | 26 | 23 | 25 | 23 | 23
  WT, Day 91 | 2233.9 (2.38) | 2606.6 (2.43) | 5793.7 (2.76) | 3917.9 (2.55) | 8607.5 (2.42) | 4050.6 (2.41) | 6861.6 (2.71)
  WT, Day 181: number analyzed (Participants) | 8 | 14 | 24 | 21 | 22 | 23 | 22
  WT, Day 181 | 2662.1 (2.42) | 2105.0 (2.39) | 3138.8 (2.68) | 2088.1 (3.33) | 4413.8 (1.98) | 2126.5 (2.64) | 3018.1 (3.28)
  Omicron BA.1, Day 1 | 399.6 (8.15) | 545.1 (4.46) | 500.0 (4.83) | 188.7 (5.86) | 410.2 (4.91) | 366.8 (5.77) | 445.8 (5.20)
  Omicron BA.1, Day 15: number analyzed (Participants) | 13 | 14 | 27 | 27 | 25 | 24 | 24
  Omicron BA.1, Day 15 | 2357.5 (2.88) | 2723.1 (2.28) | 4770.9 (3.28) | 2180.5 (3.27) | 4997.7 (2.76) | 4767.7 (2.05) | 10237.9 (2.73)
  Omicron BA.1, Day 29: number analyzed (Participants) | 13 | 14 | 27 | 26 | 26 | 26 | 21
  Omicron BA.1, Day 29 | 2317.0 (3.16) | 2270.5 (2.62) | 4263.8 (3.37) | 1876.5 (3.48) | 4395.3 (2.54) | 3859.4 (2.43) | 7582.7 (2.98)
  Omicron BA.1, Day 91: number analyzed (Participants) | 10 | 14 | 26 | 23 | 25 | 23 | 23
  Omicron BA.1, Day 91 | 2207.8 (2.56) | 2536.0 (3.11) | 2864.4 (3.58) | 1619.9 (3.60) | 3244.6 (3.70) | 2009.2 (2.79) | 3410.5 (2.80)
  Omicron BA.1, Day 181: number analyzed (Participants) | 8 | 14 | 24 | 21 | 22 | 23 | 22
  Omicron BA.1, Day 181 | 1568.7 (2.96) | 2070.4 (2.78) | 1832.4 (3.63) | 1004.8 (4.54) | 1647.4 (2.59) | 1401.6 (3.35) | 2040.9 (4.05)
  Omicron BA.2, Day 1 | 435.6 (7.06) | 497.7 (4.14) | 503.5 (5.36) | 205.4 (5.13) | 513.1 (5.14) | 432.5 (6.49) | 527.6 (5.47)
  Omicron BA.2, Day 15: number analyzed (Participants) | 13 | 14 | 27 | 27 | 25 | 24 | 24
  Omicron BA.2, Day 15 | 2262.6 (3.03) | 2643.6 (2.14) | 5348.4 (3.24) | 2383.0 (2.77) | 5587.0 (2.89) | 5046.6 (2.01) | 7229.7 (4.90)
  Omicron BA.2, Day 29: number analyzed (Participants) | 13 | 14 | 27 | 26 | 26 | 26 | 21
  Omicron BA.2, Day 29 | 1426.0 (3.24) | 2128.8 (2.16) | 4590.7 (3.15) | 2134.2 (2.84) | 5148.6 (3.02) | 3364.4 (2.55) | 7440.6 (2.99)
  Omicron BA.2, Day 91: number analyzed (Participants) | 10 | 14 | 26 | 23 | 25 | 23 | 23
  Omicron BA.2, Day 91 | 1672.7 (2.43) | 1580.6 (2.49) | 2430.5 (3.25) | 1399.4 (3.06) | 2931.6 (3.16) | 1723.1 (2.68) | 3094.9 (2.76)
  Omicron BA.2, Day 181: number analyzed (Participants) | 8 | 14 | 24 | 21 | 22 | 23 | 22
  Omicron BA.2, Day 181 | 1525.3 (3.56) | 1359.2 (2.45) | 1362.4 (4.18) | 903.8 (3.81) | 1801.2 (2.74) | 1151.5 (3.23) | 1823.2 (3.56)
  Omicron BA.5, Day 1 | 263.2 (7.74) | 374.9 (5.04) | 254.4 (6.17) | 100.0 (5.24) | 276.8 (5.69) | 253.6 (5.89) | 381.9 (5.21)
  Omicron BA.5, Day 15: number analyzed (Participants) | 13 | 14 | 27 | 27 | 25 | 24 | 24
  Omicron BA.5, Day 15 | 1336.7 (2.87) | 1442.8 (2.04) | 1985.9 (3.05) | 1017.1 (3.13) | 2756.7 (3.26) | 2354.2 (2.79) | 5956.0 (3.27)
  Omicron BA.5, Day 29: number analyzed (Participants) | 13 | 14 | 27 | 26 | 26 | 26 | 21
  Omicron BA.5, Day 29 | 1213.4 (3.28) | 1364.1 (1.97) | 1613.8 (3.47) | 832.2 (3.01) | 2304.2 (3.27) | 1532.3 (2.91) | 4310.4 (3.37)
  Omicron BA.5, Day 91: number analyzed (Participants) | 10 | 14 | 26 | 23 | 25 | 23 | 23
  Omicron BA.5, Day 91 | 1024.5 (2.63) | 1072.0 (2.21) | 1027.9 (4.06) | 618.5 (3.37) | 1341.2 (3.93) | 1002.9 (3.58) | 1923.5 (3.17)
  Omicron BA.5, Day 181: number analyzed (Participants) | 8 | 14 | 24 | 21 | 22 | 23 | 22
  Omicron BA.5, Day 181 | 928.1 (4.27) | 908.0 (2.05) | 822.1 (4.54) | 383.7 (4.74) | 957.2 (3.49) | 483.9 (4.56) | 1108.4 (4.33)
  Delta, Day 1 | 496.3 (5.55) | 494.9 (3.73) | 587.7 (4.46) | 249.4 (3.78) | 591.6 (3.53) | 474.0 (5.12) | 500.2 (5.21)
  Delta, Day 15: number analyzed (Participants) | 13 | 14 | 27 | 27 | 25 | 24 | 24
  Delta, Day 15 | 1584.4 (2.84) | 1907.8 (2.38) | 3478.6 (2.59) | 2066.0 (2.28) | 4606.8 (2.32) | 3455.8 (2.24) | 9241.4 (2.55)
  Delta, Day 29: number analyzed (Participants) | 13 | 14 | 27 | 26 | 26 | 26 | 21
  Delta, Day 29 | 1449.8 (2.70) | 1641.1 (2.74) | 3253.1 (2.75) | 1865.1 (2.49) | 3810.1 (2.33) | 3295.5 (2.36) | 5906.9 (2.66)
  Delta, Day 91: number analyzed (Participants) | 10 | 14 | 26 | 23 | 25 | 23 | 23
  Delta, Day 91 | 1200.2 (2.58) | 1212.4 (3.33) | 2020.3 (3.87) | 1249.9 (2.94) | 2627.1 (2.72) | 1685.9 (2.87) | 2393.6 (2.71)
  Delta, Day 181: number analyzed (Participants) | 8 | 14 | 24 | 21 | 22 | 23 | 22
  Delta, Day 181 | 1210.5 (2.84) | 1064.9 (2.99) | 1300.1 (3.16) | 896.5 (2.93) | 1482.6 (2.20) | 841.7 (2.93) | 1277.6 (3.37)

8. Secondary Outcome: Geometric Mean Increase (GMI) From Baseline of Neutralizing Ab Titers Against Pseudovirus Bearing S Protein From SARS-CoV-2 WT, Omicron, and Delta Variants at Each Collection Time Point
Time Frame: At Day 15, Day 29, Day 91, and Day 181
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: Fold increase
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg)
Number analyzed (Participants) | 13 | 14 | 27 | 27 | 26 | 26 | 24
Fold increase
  Wild Type (WT), Day 15: number analyzed (Participants) | 13 | 14 | 27 | 27 | 25 | 24 | 24
  Wild Type (WT), Day 15 | 2.14 (2.500) | 3.16 (2.765) | 4.10 (2.687) | 5.25 (3.292) | 4.89 (3.329) | 8.10 (3.171) | 13.31 (4.397)
  WT, Day 29: number analyzed (Participants) | 13 | 14 | 27 | 26 | 26 | 26 | 21
  WT, Day 29 | 1.89 (2.337) | 2.48 (2.934) | 3.47 (2.557) | 7.16 (2.456) | 7.20 (3.118) | 6.86 (3.792) | 11.74 (3.453)
  WT, Day 91: number analyzed (Participants) | 10 | 14 | 26 | 23 | 25 | 23 | 23
  WT, Day 91 | 1.06 (1.938) | 2.25 (2.948) | 3.28 (2.709) | 4.83 (2.721) | 4.42 (2.883) | 3.61 (2.792) | 4.14 (2.928)
  WT, Day 181: number analyzed (Participants) | 8 | 14 | 24 | 21 | 22 | 23 | 22
  WT, Day 181 | 1.02 (2.201) | 1.83 (2.917) | 1.82 (3.000) | 2.79 (2.204) | 1.86 (2.586) | 1.98 (2.636) | 1.83 (3.615)
  Omicron BA.1, Day 15: number analyzed (Participants) | 13 | 14 | 27 | 27 | 25 | 24 | 24
  Omicron BA.1, Day 15 | 3.72 (3.328) | 5.00 (5.923) | 8.64 (3.575) | 11.56 (3.789) | 12.04 (3.518) | 11.09 (4.294) | 23.51 (4.705)
  Omicron BA.1, Day 29: number analyzed (Participants) | 13 | 14 | 27 | 26 | 26 | 26 | 21
  Omicron BA.1, Day 29 | 3.66 (2.794) | 4.17 (6.567) | 7.71 (3.348) | 10.54 (3.314) | 11.12 (3.793) | 11.05 (3.888) | 20.89 (4.123)
  Omicron BA.1, Day 91: number analyzed (Participants) | 10 | 14 | 26 | 23 | 25 | 23 | 23
  Omicron BA.1, Day 91 | 2.37 (2.675) | 4.64 (7.041) | 5.31 (3.180) | 8.94 (3.448) | 7.76 (3.798) | 6.55 (3.411) | 7.39 (3.460)
  Omicron BA.1, Day 181: number analyzed (Participants) | 8 | 14 | 24 | 21 | 22 | 23 | 22
  Omicron BA.1, Day 181 | 1.39 (2.863) | 3.81 (6.801) | 3.40 (3.165) | 6.30 (3.695) | 3.22 (3.122) | 4.27 (3.411) | 4.38 (4.698)
  Omicron BA.2, Day 15: number analyzed (Participants) | 13 | 14 | 27 | 27 | 25 | 24 | 24
  Omicron BA.2, Day 15 | 3.64 (3.177) | 5.31 (5.736) | 9.50 (3.567) | 11.63 (3.182) | 10.51 (3.586) | 9.77 (4.246) | 13.44 (6.178)
  Omicron BA.2, Day 29: number analyzed (Participants) | 13 | 14 | 27 | 26 | 26 | 26 | 21
  Omicron BA.2, Day 29 | 2.30 (3.466) | 4.27 (5.859) | 8.16 (3.503) | 10.80 (3.391) | 10.59 (3.758) | 8.00 (5.258) | 16.01 (4.056)
  Omicron BA.2, Day 91: number analyzed (Participants) | 10 | 14 | 26 | 23 | 25 | 23 | 23
  Omicron BA.2, Day 91 | 1.81 (2.668) | 3.17 (6.083) | 4.52 (3.098) | 6.88 (3.823) | 5.44 (3.831) | 4.76 (4.024) | 5.48 (3.018)
  Omicron BA.2, Day 181: number analyzed (Participants) | 8 | 14 | 24 | 21 | 22 | 23 | 22
  Omicron BA.2, Day 181 | 1.30 (2.624) | 2.73 (5.862) | 2.57 (4.061) | 4.96 (2.984) | 2.77 (3.565) | 2.90 (3.669) | 3.06 (4.172)
  Omicron BA.5, Day 15: number analyzed (Participants) | 13 | 14 | 27 | 27 | 25 | 24 | 24
  Omicron BA.5, Day 15 | 3.64 (3.370) | 3.85 (6.017) | 6.94 (3.677) | 10.16 (3.210) | 9.57 (3.709) | 7.86 (3.871) | 15.67 (3.821)
  Omicron BA.5, Day 29: number analyzed (Participants) | 13 | 14 | 27 | 26 | 26 | 26 | 21
  Omicron BA.5, Day 29 | 3.30 (3.031) | 3.63 (5.877) | 5.64 (3.458) | 8.72 (3.011) | 8.99 (3.658) | 5.93 (3.645) | 12.69 (3.418)
  Omicron BA.5, Day 91: number analyzed (Participants) | 10 | 14 | 26 | 23 | 25 | 23 | 23
  Omicron BA.5, Day 91 | 1.93 (3.136) | 2.87 (6.515) | 3.78 (3.451) | 5.94 (2.791) | 4.55 (3.842) | 4.03 (2.932) | 4.60 (2.654)
  Omicron BA.5, Day 181: number analyzed (Participants) | 8 | 14 | 24 | 21 | 22 | 23 | 22
  Omicron BA.5, Day 181 | 1.25 (2.678) | 2.42 (6.001) | 3.14 (3.293) | 4.16 (2.728) | 2.75 (3.822) | 2.13 (2.808) | 2.62 (3.846)
  Delta, Day 15: number analyzed (Participants) | 13 | 14 | 27 | 27 | 25 | 24 | 24
  Delta, Day 15 | 2.32 (2.100) | 3.86 (3.575) | 5.50 (3.041) | 8.28 (2.837) | 7.23 (3.225) | 6.27 (3.502) | 18.44 (5.067)
  Delta, Day 29: number analyzed (Participants) | 13 | 14 | 27 | 26 | 26 | 26 | 21
  Delta, Day 29 | 2.12 (2.002) | 3.31 (3.919) | 5.16 (2.783) | 7.76 (2.982) | 6.73 (3.424) | 7.12 (3.677) | 13.62 (4.023)
  Delta, Day 91: number analyzed (Participants) | 10 | 14 | 26 | 23 | 25 | 23 | 23
  Delta, Day 91 | 1.26 (1.717) | 2.45 (3.973) | 3.26 (2.973) | 5.27 (2.817) | 4.12 (3.235) | 4.16 (3.198) | 4.41 (3.020)
  Delta, Day 181: number analyzed (Participants) | 8 | 14 | 24 | 21 | 22 | 23 | 22
  Delta, Day 181 | 0.97 (2.131) | 2.15 (3.829) | 2.16 (3.188) | 4.14 (2.414) | 1.96 (3.087) | 2.10 (2.982) | 2.37 (3.394)

9. Secondary Outcome: Percentage of Participants With Neutralizing Seroresponse of Serum SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 Variants Specific Ab at Day 29
Description: Seroresponse was defined as post-boost titers >= 4 times pre-boost (baseline) titers for participants with titer >= LLOQ at pre-vaccination and as post-booster titer >= 4 times LLOQ for participants with titer < LLOQ at pre vaccination.
Time Frame: At day 29 (28 days after the booster dose)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg)
Number analyzed (Participants) | 13 | 14 | 27 | 26 | 26 | 26 | 21
Percentage of participants
  Ancestral WT | 15.4 [1.9 to 45.4] | 21.4 [4.7 to 50.8] | 33.3 [16.5 to 54.0] | 69.2 [48.2 to 85.7] | 69.2 [48.2 to 85.7] | 50.0 [29.9 to 70.1] | 76.2 [52.8 to 91.8]
  Omicron BA.1 | 38.5 [13.9 to 68.4] | 21.4 [4.7 to 50.8] | 74.1 [53.7 to 88.9] | 65.4 [44.3 to 82.8] | 84.6 [65.1 to 95.6] | 76.9 [56.4 to 91.0] | 95.2 [76.2 to 99.9]
  Omicron BA.2 | 30.8 [9.1 to 61.4] | 28.6 [8.4 to 58.1] | 77.8 [57.7 to 91.4] | 73.1 [52.2 to 88.4] | 73.1 [52.2 to 88.4] | 61.5 [40.6 to 79.8] | 90.5 [69.9 to 98.8]
  Omicron BA.5 | 38.5 [13.9 to 68.4] | 28.6 [8.4 to 58.1] | 48.1 [28.7 to 68.1] | 73.1 [52.2 to 88.4] | 73.1 [52.2 to 88.4] | 50.0 [29.9 to 70.1] | 81.0 [58.1 to 95.6]

10. Primary Outcome: Number of Participants With Each Abnormal Clinical Safety Laboratory Finding for 8 Days After Study Vaccination
Description: An abnormal laboratory is defined as any value outside of the normal range. Normal ranges were: Alanine Aminotransferase: (Female: 10-32 micro (u)/ liter (L); Male: 10-40 u/L); Alkaline Phosphatase: (Female: 30-115 u/L; Male: 43-115 u/L); Aspartate Aminotransferase: (Female: 10-36 u/L; Male: 10-43 u/L); Bilirubin total: 0.1-1.1 milligram (mg)/deciliter (dL); Bilirubin, Direct: 0-0.4 mg/dL ;Creatinine:0.7-1.4 mg/dL; Eosinophils: 0%-7%; Eosinophils/Leukocytes: 0.00-0.80 x 10^3/uL ; Erythrocytes: (Female: 3.70-5.20 x 10^6/uL; Male: 4.63-6.08x 10^6/uL); Hemoglobin: (Female: 11.0-15.5 gram (g)/dL; Male: 12.5-17.0 g/dL); Leukocytes: 3.70-11.00 x 10^3/uL; Lymphocytes 12.0%-46.0%; Lymphocytes/Leukocytes: 0.90-3.60 x 10^3/uL; Monocytes/Leukocytes: 0.00-1.20 x 10^3/uL; Neutrophils: 4.0% - 71.0%; Neutrophils/Leukocytes:1.70-7.90x 10^3/uL; Platelets: 163-375 x 10^3/uL; Urea Nitrogen: 5-20 mg/dL.
Time Frame: 8 days from vaccination at Day 1
Population: Analysis was performed on the Safety set who received 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg)
Number analyzed (Participants) | 15 | 15 | 30 | 30 | 30 | 30 | 30
Participants
  Alanine Aminotransferase (High) | 0 | 0 | 1 | 1 | 6 | 1 | 3
  Alanine Aminotransferase (Low) | 0 | 0 | 4 | 2 | 1 | 1 | 2
  Alkaline Phosphatase (High) | 0 | 0 | 1 | 0 | 1 | 2 | 2
  Aspartate Aminotransferase (High) | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Bilirubin (High) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Creatinine (High) | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Eosinophils (High) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils/Leukocytes (High) | 2 | 1 | 1 | 1 | 0 | 1 | 1
  Erythrocytes (High) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Erythrocytes (Low) | 4 | 0 | 1 | 3 | 8 | 5 | 8
  Hemoglobin (High) | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (Low) | 0 | 0 | 0 | 2 | 1 | 0 | 1
  Leukocytes (High) | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Leukocytes (Low) | 1 | 0 | 0 | 0 | 3 | 0 | 1
  Lymphocytes (High) | 2 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes/Leukocytes (High) | 2 | 2 | 2 | 3 | 2 | 3 | 3
  Monocytes/Leukocytes (High) | 0 | 1 | 2 | 2 | 2 | 0 | 0
  Neutrophils (High) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophils (Low) | 1 | 1 | 2 | 1 | 3 | 1 | 0
  Neutrophils/Leukocytes (High) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Neutrophils/Leukocytes (Low) | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Platelets (High) | 3 | 5 | 0 | 2 | 1 | 0 | 0
  Platelets (Low) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urea Nitrogen (High) | 0 | 0 | 0 | 1 | 1 | 3 | 2

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs), Medically Attended Adverse Events (MAAEs), and Adverse Events of Special Interest (AESIs) were collected through the entire period of the study (from Day 1 up to study end [Day 180]). Solicited adverse events were collected from Day 1-7. Unsolicited adverse events from Day 1-28. Abnormal Clinical Safety Laboratory Findings from Day 1-8. Non-Serious Covid-19 Adverse Events from Day 1 up to Study End [Day 180] after Study Vaccination.
Description: Adverse events were assessed in safety set which included all participants that received the study intervention administration.
Arm/Group | Part B: CV0501 Dose Cohort 6 (3 μg) | Part B: CV0501 Dose Cohort 7 (6 μg) | Part A: CV0501 Dose Cohort 1 (12 μg) | Part A: CV0501 Dose Cohort 2 (25 μg) | Part A: CV0501 Dose Cohort 3 (50 μg) | Part A: CV0501 Dose Cohort 4 (100 μg) | Part A: CV0501 Dose Cohort 5 (200 μg)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/30 | 0/30 | 1/30 | 2/30 | 0/30
Other Adverse Events (participants affected / at risk) | 11/15 | 10/15 | 18/30 | 22/30 | 19/30 | 22/30 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part B: CV0501 Dose Cohort 6 (3 μg) (N=15) | Part B: CV0501 Dose Cohort 7 (6 μg) (N=15) | Part A: CV0501 Dose Cohort 1 (12 μg) (N=30) | Part A: CV0501 Dose Cohort 2 (25 μg) (N=30) | Part A: CV0501 Dose Cohort 3 (50 μg) (N=30) | Part A: CV0501 Dose Cohort 4 (100 μg) (N=30) | Part A: CV0501 Dose Cohort 5 (200 μg) (N=30)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part B: CV0501 Dose Cohort 6 (3 μg) (N=15) | Part B: CV0501 Dose Cohort 7 (6 μg) (N=15) | Part A: CV0501 Dose Cohort 1 (12 μg) (N=30) | Part A: CV0501 Dose Cohort 2 (25 μg) (N=30) | Part A: CV0501 Dose Cohort 3 (50 μg) (N=30) | Part A: CV0501 Dose Cohort 4 (100 μg) (N=30) | Part A: CV0501 Dose Cohort 5 (200 μg) (N=30)
Injection site pain (General disorders) | 5 (5) | 9 (9) | 14 (14) | 19 (19) | 15 (15) | 19 (19) | 22 (22)
Fatigue (General disorders) | 1 (1) | 0 (0) | 5 (5) | 14 (14) | 10 (10) | 15 (16) | 14 (14)
Chills (General disorders) | 1 (1) | 0 (0) | 3 (3) | 5 (5) | 3 (3) | 11 (11) | 11 (11)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 9 (10)
Injection site swelling (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 6 (6)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Administration site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 8 (8) | 10 (10) | 10 (10) | 16 (16) | 17 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 3 (3) | 6 (6) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 4 (4) | 5 (5) | 9 (9) | 9 (9) | 13 (13) | 13 (13)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 4 (4) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 5 (5) | 4 (4) | 6 (6)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT05477186/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT05477186/SAP_001.pdf